CLINICAL TRIAL: NCT00789243
Title: The Effect of Ischaemic-Reperfusion and Ischaemic Preconditioning on the Endogenous Fibrinolysis in Man
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: University of Aarhus (Other); University of Oxford (Other)
Responsible Party: Christian M Pedersen, clinical research fellow, University of Edinburgh
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CMP 2
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-10

CONDITIONS: Ischaemic Heart Diseases
Keywords: Ischaemia reperfusion; t-PA; Fibrinolysis; Endothelial function; Local and remote ischaemic preconditioning
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Prior to 20 mins of ischaemia induced by a blood pressure cuff inflated to 200 mmHg around the upper non-dominant arm, local ischaemic preconditioning will be induced by inflating a cuff around the non-dominant arm to 200 mmHg for 5 mins followed by 5 mins of reperfusion. This cycle will be repeated 3 times.
  Interventions: Procedure: Forearm vascular study
- 2 (Active Comparator): Prior to 20 mins of ischaemia induced by a blood pressure cuff inflated to 200 mmHg around the upper non-dominant arm, remote ischaemic preconditioning will be induced by inflating a cuff around the dominant arm to 200 mmHg for 5 mins followed by 5 mins of reperfusion. This cycle will be repeated 3 times.
  Interventions: Procedure: Forearm vascular study
- 3 (Placebo Comparator): Prior to 20 mins of ischaemia induced by a blood pressure cuff inflated to 200 mmHg around the upper non-dominant arm, sham will be performed by inflating a cuff to 10 mmHg for 5 mins followed by 5 mins of deflation. This cycle will be repeated 3 times.
  Interventions: Procedure: Forearm vascular study

INTERVENTIONS:
Procedure: Forearm vascular study — Forearm blood flow measured by venous occlusion plethysmography during interarterial infusion of substance P (2,4,8 pmol/min). Venous blood sampling via cannula in antecubital fossa.

SUMMARY:
Heart attacks are usually caused by a blood clot blocking an artery supplying blood to the heart. Current treatments are designed at relieving this blockage as quickly as possible to minimise damage to the heart muscle. However in restoring the supply of blood local damage known as "ischaemia-reperfusion injury" may occur. The aim of this study is to assess how clot forming and clot dissolving pathways are affected during this process, and examine the role of a natural inflammatory hormone, bradykinin. This will help us to understand the mechanism by which ischaemia-reperfusion injury may occur and to devise new treatments for heart attacks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males between 18-65 years of ages, non-smokers.

Exclusion Criteria:

* Any concurrent illness or chronic medical condition. Concurrent use of vasoactive medication. Smoking history.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Net t-PA release from the endothelium after ischaemia reperfusion and ischaemic preconditioning | Throughout the study

SECONDARY OUTCOMES:
Change in forearm blood flow after ischaemia reperfusion and ischaemic preconditioning | throughout the study
Change in platelet-monocyte-binding after ischaemia reperfusion and ischaemic preconditioning | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, PhD, FRCP, Study Director — University of Edinburgh; Rajesh K Kharbanda, PhD, FRCP, Study Director — University of Oxford
Locations (1):
- University of Edinburgh, 49 Little France Crescent, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Pedersen CM, Barnes G, Schmidt MR, Botker HE, Kharbanda RK, Newby DE, Cruden NL. Ischaemia-reperfusion injury impairs tissue plasminogen activator release in man. Eur Heart J. 2012 Aug;33(15):1920-7. doi: 10.1093/eurheartj/ehr380. Epub 2011 Oct 11. PMID 21990263
- [Derived] Pedersen CM, Cruden NL, Schmidt MR, Lau C, Botker HE, Kharbanda RK, Newby DE. Remote ischemic preconditioning prevents systemic platelet activation associated with ischemia-reperfusion injury in humans. J Thromb Haemost. 2011 Feb;9(2):404-7. doi: 10.1111/j.1538-7836.2010.04142.x. No abstract available. PMID 21083644